CLINICAL TRIAL: NCT02305992
Title: Effect of Sympathetic Blockade on the Success and Survival of Arteriovenous Fistula
Brief Title: Regional Anesthesia for Arteriovenous Fistula
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Looking for funding opportunities
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-123
Record Dates: First submitted 2014-11-11; First posted 2014-12-03 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Axillary Block with 0.5% Ropivicaine (Experimental): Patients will receive an axillary block using an ultrasound-guided technique. After skin infiltration with 1 mL of 2% lidocaine, a 22-gauge insulated needle is advanced in-plane from the cephalic aspect of the transducer toward the posterior aspect of the axillary artery. Prior to injection, the syringe is aspirated to confirm extra-vascular placement of the needle. 20 mL solution of 0.5% ropivicaine is then injected slowly, with syringe aspiration after every 5 mL injection to confirm extravascular placement.
  Interventions: Procedure: Axillary Block with 0.5% Ropivicaine
- Stellate Ganglion Block with 0.2% Ropivicaine (Experimental): Patients will receive stellate ganglion block and local anesthetic using an ultrasound-guided technique.After skin infiltration with 1 mL of 2% lidocaine, a 22-gauge insulated needle is advanced in-plane from the lateral position toward the anterior aspect of longus colli muscle just posterior to the internal jugular vein. Prior to injection, the syringe is aspirated to confirm extra-vascular placement of the needle. 10 mL of 0.2% ropivicaine is then injected slowly, with syringe aspiration after every 5 mL injection to confirm extravascular placement.
  Interventions: Procedure: Stellate ganglion block with 0.2% Ropivicaine
- Local anesthetic infiltration with 0.25% Bupivicaine (Active Comparator): Patients will receive local anesthetic infiltration of 0.25% Bupivicaine at the surgical site which will last approximately 6 hours.
  Interventions: Procedure: Local anesthetic infiltration with 0.25% Bupivicaine

INTERVENTIONS:
Procedure: Axillary Block with 0.5% Ropivicaine — Axillary blocks are regional anesthesia techniques that are sometimes employed as an alternative to general anesthesia for surgery of the shoulder, arm, forearm, wrist and hand. In this case, ultra-sound technique will be used.
  Arms: Axillary Block with 0.5% Ropivicaine
Procedure: Stellate ganglion block with 0.2% Ropivicaine — A stellate ganglion block is an injection of local anesthetic in the sympathetic nerve tissue of the neck. These nerves are a part of the sympathetic nervous system. The nerves are located on either side of the voice box, in the neck
  Arms: Stellate Ganglion Block with 0.2% Ropivicaine
Procedure: Local anesthetic infiltration with 0.25% Bupivicaine — Patients will receive local anesthetic infiltration of 0.25% Bupivicaine at the surgical site which will last approximately 6 hours.
  Arms: Local anesthetic infiltration with 0.25% Bupivicaine

SUMMARY:
Once kidney function goes below 10 to 15 percent of normal, dialysis treatments or a kidney transplant are necessary to sustain life. One type of dialysis is hemodialysis which cleans blood by removing it from the body and passing it through a dialyzer, or artificial kidney. To maximize the amount of blood cleansed during hemodialysis treatments, there should be continuous high volumes of blood flow. A fistula used for hemodialysis is a direct connection of an artery to a vein. Once an arteriovenous fistula (AVF) is created it is a natural part of the body. This is the preferred type of access because once the fistula properly matures and gets bigger and stronger; it provides an access with good blood flow that can last for decades. After the fistula is surgically created, it can take weeks to months before the fistula matures and is ready to be used for hemodialysis. There have been surgical factors identified; one of them being the anesthetic used which may cause a fistula not to survive. This study will look at comparing 3 anesthetic techniques: axillary block (AB) versus stellate ganglion (SGB) block+local anesthetic versus local anesthetic (LA).

DETAILED DESCRIPTION:
To allow for chronic hemodialysis (HD), patients with end-stage renal disease (ESRD) require permanent vascular access in the form of either arteriovenous graft (AVG) or arteriovenous fistula (AVF). The latter option is the preferred form of vascular access given the lower rate of thrombosis, fewer interventions required, longer survival for vascular access and lower rate of infection as compared to AVG (1). Despite this, earlier reports have suggested that the initial failure rate of AVF approximates to 25% (2). A permanent vascular access is considered adequate when it has sufficient size (i.e. greater than 0.6 cm) for easy cannulation and a flow rate of approximately 600 mL/min for dialysis (1, 3). However, postoperative AVF blood flow may be compromised by arterial vasospasm and sympathetic activity from surgical manipulations (4, 5). Inadequate flow rate in the postoperative period can result in early thrombus formation at the fistula and, if left untreated, can lead to permanent loss of vascular access(6). Over the years, researchers have identified a number of patient and surgical factors that may influence the success and long-term survival of AVF, and recent evidence suggests that the choice of anesthetic techniques may play a significant role (7).

Vascular access surgery is usually conducted under either a) general anesthesia (GA), b) local anesthetics (LA) infiltrations with sedations, or c) regional anesthesia in the form of brachial plexus block (BPB). GA, while providing both anesthesia and analgesia, can present a challenge for maintaining intraoperative hemodynamic stability as patients with ESRD often have other significant comorbidities. LA infiltrations, though offering simplicity, does not provide motor blockade and patient movement can be a surgical challenge. LA requires multiple injections during the case. BPB thus presents as an attractive option as it provides both dense and prolonged sensory and motor blockade while avoiding the cardiopulmonary stress imposed by GA. Additionally, the sympathectomy associated with BPB has been shown to improve postoperative AVF blood flow through decreasing peripheral vascular resistance and increasing vasodilation and blood flow velocity (8-11). Similarly, stellate ganglion block (SGB), which offers sympathetic blockade without analgesic effect, has also been shown to augment postoperative AVF blood flow and average peak flow velocity and shorten maturation time when combined with LA infiltrations (5, 12).

Though it has been shown that regional anesthesia can affect a number of physiological parameters following AVF formation, it is not yet clear how fistula survival can be affected by the modification of these parameters. The investigators conducted a literature search in July 2013 using MEDLINE database. Two key words, one from List A and one from List B, were joined with the term "and" in all possible combinations for the literature search. Key words from List A included "arteriovenous fistula", "AVF", "vascular access", "dialysis", and "dialysis access". List B included "regional anesthesia", "brachial plexus block," "BPB", "brachial plexus", "stellate ganglion", "SGB", "sympathectomy", "supraclavicular", "infraclavicular", "axillary", and "interscalene". Search results were limited to English articles only. Abstracts were not included in the search results. To the investigators knowledge, no randomized trial has been conducted to directly compare the effect of axillary block (AB) against LA infiltration with or without SGB on AVF success in patients with ESRD. This will be the primary objective of the investigators study. To do so, the investigators intend to conduct a prospective randomized controlled trial at a tertiary vascular surgical center in Hamilton.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ESRD undergoing radio-cephalic AVF

Exclusion Criteria:

* Previous AVF procedures
* significant stenosis (>50% diameter reduction)
* calcifications of radial artery or cephalic vein
* radial artery diameter <1.6mm
* cephalic vein diameter <2.0mm
* history of pre-existing unilateral recurrent laryngeal nerve palsy
* pre-existing unilateral phrenic nerve palsy
* coagulopathy or pre-existing conditions that require anticoagulants or anti-platelet therapies
* history of IV drug use
* documented allergic reactions to local anesthetics
* pregnancy
* morbid obesity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Arteriovenous fistula flow | 1 hour post-operatively
  Arteriovenous fistula in mL/min

SECONDARY OUTCOMES:
Change in limb temperature pre-anesthetic and post-anesthetics | 1 hour post-operatively
Duration of intraoperative procedure | 3 hours post-operatively
Rate of conversion to general anesthetic | 1 day post-operatively
Anesthesia-related adverse events | 1 day post-operatively
Maturation time | 2 months post-operatively
Patient Satisfaction | 2 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Turlough O'Hare, MD, Principal Investigator — St. Joseph's Healthcare Hamilton/McMaster Univeristy
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Allon M, Robbin ML. Increasing arteriovenous fistulas in hemodialysis patients: problems and solutions. Kidney Int. 2002 Oct;62(4):1109-24. doi: 10.1111/j.1523-1755.2002.kid551.x. PMID 12234281
- [Background] He GW, Yang CQ. Radial artery has higher receptor-mediated contractility but similar endothelial function compared with mammary artery. Ann Thorac Surg. 1997 May;63(5):1346-52. doi: 10.1016/s0003-4975(97)00106-9. PMID 9146326
- [Background] Fries A. [Environmental access to a rehabilitation center as a determinant of attitude to handicapped persons? A comparative empirical study of assumptions of the "contact hypothesis"]. Rehabilitation (Stuttg). 1991 Feb;30(1):28-37. German. PMID 1828300